CLINICAL TRIAL: NCT06460558
Title: "Impact of an Automated Closed-loop Insulin Infusion System on Adherence to Physical Activity in Patients With Type 1 Diabetes "
Brief Title: T1D Closed-loop and Physical Activity
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24Endocrino01
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Diabetes type1
MeSH Terms: interventions — Insulin Infusion Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 diabetes with insulin infusion system
  Interventions: Other: Type 1 diabetes with insulin infusion system

INTERVENTIONS:
Other: Type 1 diabetes with insulin infusion system — No intervention
  Other Names: No intervention

SUMMARY:
"Physical activity is recognized as beneficial for patients living with type 1 diabetes (T1DM), with a demonstrated effect not only on HbA1c control [1] but also on reducing the incidence of diabetes-related complications [2,3]. It is recommended that patients living with T1DM perform 150 minutes of accumulated physical activity per week, without exceeding two consecutive days without physical activity [4]. Indeed, one meta-analysis reported that moderately vigorous activity (≥4.5 METs) was beneficial compared with lower-intensity activity, while three other studies noted that only vigorous physical activity (≥6 METs) predicted lower all-cause mortality rates [5]. However, T1DM can represent a major obstacle to physical activity because of the occurrence of fairly frequent hypoglycemia, including after physical effort, the need for early resugaring but also the risk of hyperglycemia (rebound or with certain activities) [6]. The advent of automated insulin delivery systems has led to a significant improvement in time on target and a reduction in the frequency of hypoglycemia, including during physical activity in some studies [7-9]. The aim of this study is therefore to evaluate, in a cohort of patients with T1DM, whether the implementation of a closed-loop automated insulin delivery system increases physical activity in patients with T1DM. Based on the interpretation of the ONAPS-PAQ [10], the investigator hypothesize that the implementation of the closed-loop system enables an individual to reach the 3000 MET/min/week threshold (considered ""Active+"" from this threshold onwards).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes defined by clinical history and positive measurement of autoantibodies (anti-GAD or IA2), evolving for more than 6 months and treated by insulin pump for at least 6 months, for whom an indication for automated insulin delivery is retained, by criteria of glycemic control (HbA1c ≥ 8% and/or significant glycemic variability and/or severe hypoglycemia) or poor quality of life, in accordance with reimbursement criteria validated by the CNAM for available systems.
* For women, existence of effective contraception (hormonal or mechanical) and no plans for pregnancy during the study period.
* Having a Health Care insurance."" "

Exclusion Criteria:

* Patient already involved in another experimental study
* Patient in a particular situation deemed incompatible with the study by the investigator
* Patient living in a department other than Alpes-Maritimes or Var
* Pregnant women
* Presence of a contraindication to physical activity
* Patient with linguistic or psychological incapacity to understand written information
* Patient refusing to give consent
* Patient deprived of liberty by administrative or judicial decision, under guardianship or trusteeship"" "

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Selection visit - Patients with T1DM referred to Nice University Hospital are offered the opportunity to take part in the study without obligation (D0).
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-11-06 (Estimated); Study Completion 2026-05-06 (Estimated)

PRIMARY OUTCOMES:
IPAQ score | At the inclusion
  "Measurement of IPAQ in METs/min/week (reflects the amount of physical activity practised using a validated questionnaire). There are seven items whose the result corresponds to the sum of the given figures. "

SECONDARY OUTCOMES:
BAPAD-1 score " | At the inclusion
  The BAPAD-1 score, validated in French, will be used to assess the usual obstacles to physical activity in T1DM. It is a Likert scale (between 0-7) composed by twelve items. Then, a mean is calculated with all the answers.
BREQ-2 | At the inclusion
  "To assess motivation to engage in physical activity, use the BREQ-2 score, validated by ONAPS. It is a Likert scale (between 0-7) composed by six items. Then, a mean is calculated with all the answers.
ONAPS PAQ | At the inclusion
  To assess sedentary behaviour, use the ONAPS PAQ score with only the sedentary behaviour section. 4 items. Then the sum of the results is calculated

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas CHEVALIER, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU NiICE, Nice, Alpes Maritimes, France